CLINICAL TRIAL: NCT00003737
Title: A Pharmacokinetic-Guided Phase II Trial of the Rebeccamycin Analog NSC# 655649 in Pediatric Patients With Relapsed/Refractory Neuroblastoma
Brief Title: Rebeccamycin Analog in Treating Children With Relapsed or Refractory Neuroblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 98-095; CDR0000066852 (Registry Identifier: PDQ (Physician Data Query)); NCI-T98-0041
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Neuroblastoma
Keywords: recurrent neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — becatecarin

INTERVENTIONS:
Drug: becatecarin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of rebeccamycin analog in treating children who have relapsed or refractory neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate to rebeccamycin analogue in children with relapsed or refractory neuroblastoma.
* Determine the toxicity of this drug in these patients.
* Identify and establish in vitro biologic correlates of clinical responses and toxicity of this drug in these patients.

OUTLINE: Patients receive rebeccamycin analogue IV over 1 hour once on days 1-5. Treatment repeats every 3 weeks for at least 2 courses in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: This study will accrue up to 30 patients within 1.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven relapsed or refractory neuroblastoma
* Measurable disease

PATIENT CHARACTERISTICS:

Age:

* Children

Performance status:

* ECOG 0-2

Life expectancy:

* At least 2 months

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin less than 1.5 mg/dL
* SGOT and SGPT less than 2.5 times upper limit of normal (ULN)
* Adequate liver function unless due to disease

Renal:

* Creatinine no greater than 1.5 times ULN OR
* Creatinine clearance at least 60 mL/min
* Adequate renal function unless due to disease

Other:

* No other serious concurrent illness
* No active uncontrolled infection
* Not pregnant
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Recovered from prior immunotherapy
* Prior autologous bone marrow transplantation allowed
* No concurrent immunotherapy

Chemotherapy:

* At least 4 weeks since prior chemotherapy and recovered
* No other concurrent systemic chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* Recovered from prior radiotherapy

Surgery:

* Not specified

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 1999-01; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Response (complete response, very good partial response, or partial response)
Freedom from progression
Time to treatment failure

SECONDARY OUTCOMES:
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Trippett, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States